CLINICAL TRIAL: NCT01907256
Title: Comparing the Aesthetic Results of Two Common Incisions in External Rhinoplasty A Randomized Trial
Brief Title: Comparing the Aesthetic Results of Two Common Incisions in External Rhinoplasty
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Tehran University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Babak Saedi, Associate professor, Tehran University of Medical Sciences
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: 92-01-48-20912
Record Dates: First submitted 2013-07-11; First posted 2013-07-24 (Estimated); Last update posted 2014-01-20 (Estimated); Status verified 2014-01

CONDITIONS: Cosmetic Outcome

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- group A (Active Comparator): stair step incisions
  Interventions: Procedure: stair step incisions
- Group B (Active Comparator): inverted V incision
  Interventions: Procedure: inverted V incision

INTERVENTIONS:
Procedure: inverted V incision — It is a type of incision
  Arms: Group B
Procedure: stair step incisions — It is a type of incision
  Arms: group A

SUMMARY:
There was not any randomize trial to show what is the best type of incision in open rhinoplasty. So, we use both self-rating by patients ,independent physician observers Visual Analogue Scale (VAS) and also a validated scar analysis to compare inverted V and stair step incisions.

DETAILED DESCRIPTION:
Approaches to rhinoplasty can be separated into two broad categories: external and endonasal, which each of them their own proponent. However, the external approach provide better exposure, critics against this technique is often due to cosmetic deformity regarding the incision. Hence, over the recent years surgeons have modified the trans-columellar incision into two big categories: gull wing and stair steps. While each of them has its own proponents, there is no randomized trial, comparing their cosmetic results.

There was not any randomize trial to show what is the best type of incision in open rhinoplasty. So, we use both self-rating by patients ,independent physician observers Visual Analogue Scale (VAS) and also a validated scar analysis to compare inverted V and stair step incisions.

ELIGIBILITY:
Inclusion Criteria:

* All patients who candidate for open rhinoplasty

Exclusion Criteria:

* Revision cases
* History of scar
* Systemic diseases

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Estimated)
Dates: Start 2012-12; Primary Completion 2013-10 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Hollunder cosmetic score | one week after surgery,
  The patients will come for office visit and their columella scars will evaluate according to above mentioned scale in one week after surgery, one month after surgery , one year after surgery
Hollunder cosmetic score | one month after surgery
  The patients will come for office visit and their columella scars will evaluate according to above mentioned scale in one week after surgery, one month after surgery , one year after surgery
Hollunder cosmetic score | one year after surgery
  The patients will come for office visit and their columella scars will evaluate according to above mentioned scale in one week after surgery, one month after surgery , one year after surgery

SECONDARY OUTCOMES:
Visual analogue score | one week after surgery,
  The patients will come for office visit and their columella scars will evaluate according to above mentioned scale inone week after surgery, one month after surgery , one year after surgery
Visual analogue score | one month after surgery
  The patients will come for office visit and their columella scars will evaluate according to above mentioned scale inone week after surgery, one month after surgery , one year after surgery
Visual analogue score | one year after surgery
  The patients will come for office visit and their columella scars will evaluate according to above mentioned scale inone week after surgery, one month after surgery , one year after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Babak Saaedi, Principal Investigator — Tehran University of Medical Sciences
Locations (1):
- Tehran University of Medical Sciences, Tehran, Tehran Province, Iran